CLINICAL TRIAL: NCT02002325
Title: THrombolysis for Acute Wake-up and Unclear-onset Strokes With Alteplase at 0.6 mg/kg Trial (THAWS)
Acronym: THAWS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Collaborators: Charitable Trust Mihara Cerebrovascular Disorder Research Promotion Fund (Unknown); Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Kazunori Toyoda, Director and Chair, Department of Cerebrovascular Medicine, National Cerebral and Cardiovascular Center, Japan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCVC-STROKE-001; UMIN000011630 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alteplase (Experimental): Intravenous tissue-type plasminogen activator (alteplase)
  Interventions: Drug: Tissue-type plasminogen activator (alteplase)
- Standard Care (Other): Standard treatment for acute stroke
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Tissue-type plasminogen activator (alteplase) — Intravenous tissue-type plasminogen activator (alteplase) 0.6mg/kg body-weight up to a maximum of 60 mg, 10% as bolus, 90% over 1 hour as infusion (plus other standard treatment if needed)
  Other Names: rt-PA; Activacin; Grtpa; Actilyse; Activase
  Arms: Alteplase
Other: Standard care — Standard treatment for acute stroke without intravenous alteplase.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to clarify efficacy and safety of MRI-based intravenous thrombolysis with alteplase for patients with acute wake-up ischemic stroke and those having acute ischemic stroke with unknown time of symptom onset.

DETAILED DESCRIPTION:
THAWS is an investigator initiated Japanese multicenter randomized controlled clinical trial of MRI based thrombolysis in patients with acute wake-up ischemic stroke and those having acute ischemic stroke with unknown time of symptom onset. Intravenous thrombolysis with alteplase of 0.6mg/kg, different from 0.9mg/kg used in other countries, is available as effective and safe treatment of acute stroke within 4.5 hours of symptom onset in Japan. However, time of symptom onset is unknown in about 25% of acute stroke patients. These patients are currently excluded from intravenous thrombolysis with alteplase. The objective of the THAWS project is to provide effective treatment options for acute stroke patients with unknown time of symptom onset. The purpose of this study is to clarify efficacy and safety of MRI-based intravenous thrombolysis with alteplase of 0.6mg/kg for patients with acute wake-up ischemic stroke and those having acute ischemic stroke with unknown time of symptom onset. Eligible patients will be selected based on MRI findings indicative of acute ischemic stroke less than 4.5 hours of age.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke with unknown symptom onset (e.g. acute wake-up ischemic stroke, acute ischemic stroke with unknown time of symptom onset)
* Last known well without neurological symptoms >4.5 hours of treatment initiation
* Treatment can be started within 4.5 hours of symptom recognition (e.g. awaking)
* Acute stroke MRI including diffusion weighted imaging (DWI) and fluid attenuated inversion recovery (FLAIR) completed
* Alberta Stroke Program Early CT score (ASPECTS) on initial DWI is 5 or more
* No marked parenchymal hyperintensity visible on FLAIR
* Initial NIHSS ≥2
* Written informed consent by patient or next of kin

Exclusion Criteria:

* Pre-stroke Modified Rankin Scale (mRS) >1 (patients who have inability to carry out all daily activities and require some help or supervision)
* Contraindications in the Japanese guideline for the intravenous application of recombinant tissue-type plasminogen activator (alteplase)

  * History of nontraumatic intracranial hemorrhage
  * History of stroke within the last 1 month (excluding transient ischemic attack)
  * History of significant head/spinal injury or surgery within the last 3 months
  * History of gastrointestinal or urinary tract bleeding within the last 21 days
  * History of major surgery or significant trauma other than head injury within the last 14 days
  * Hypersensitivity to alteplase
  * Suspected subarachnoid hemorrhage
  * Concurrent acute aortic dissection
  * Concurrent hemorrhage (e.g., intracranial, gastrointestinal, urinary tract, or retroperitoneal, hemoptysis)
  * Systolic blood pressure ≥185 mmHg despite antihypertensive therapy
  * Diastolic blood pressure ≥110 mmhg despite antihypertensive therapy
  * Significant hepatic disorder
  * Acute pancreatitis
  * Blood glucose <50mg/dL or >400 mg/dL
  * Platelet count ≤100,000/mm3
  * International normalized ratio of prothrombin time (PT-INR) >1.7 or Prolonged activated partial thromboplastin time (aPTT: >1.5 times the baseline value [>approximately 40 seconds only as a guide]) for patients on anticoagulation therapy or those with abnormal coagulation
* Any contraindication to MRI (e.g. cardiac pacemaker)
* Extensive early ischemic change in brain stem or cerebellum (e.g., more than half of brain stem or more than one hemisphere of cerebellum)
* Planned or anticipated treatment with surgery or endovascular reperfusion strategies (e.g., intra-arterial thrombolysis, mechanical recanalization techniques)
* Pregnant, lactating, or potentially pregnant
* Life expectancy 6 months or less by judgment of the investigator
* Inappropriate for study enrollment by judgment of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale 0-1 | 90 days after stroke onset

SECONDARY OUTCOMES:
Categorical shift in National Institutes of Health (NIHSS) score at 24 h | 24 hours after the initiation of treatment
Categorical shift in NIHSS score at 7 days | 7 days after the initiation of treatment
Modified Rankin Scale 0-2 | 90 days after stroke onset
Categorical shift in modified Rankin Scale score | 90 days after stroke onset
Parenchymal hemorrhage type-2 (PH-2) | 24 hours after the initiation of treatment
  MRI proven SICH
Symptomatic intracranial hemorrhage (sICH) in SITS-MOST | 24 hours after the initiation of treatment
  MRI proven SICH
sICH as defined in European Cooperative Acute Stroke Study (ECASS) II | 24 hours after the initiation of treatment
  MRI proven SICH
sICH as defined in National Institute of Neurological Disorders and Stroke (NINDS) | 24 hours after the initiation of treatment
  MRI proven SICH
Major bleeding | Up to 90 days after stroke onset
  Fatal bleeding, symptomatic bleeding in a critical area or organ, such as intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, or bleeding causing a fall in hemoglobin level of ≥2g/dL, or leading to transfusion of ≥4.5 units of whole blood or red cells according to the definition of the International Society on Thrombosis and Haemostasis
Modified Rankin Scale 6 | 90 days after stroke onset
  Death due to any cause
Infarct volume | 7 days after stroke onset
  Infarct volume on FLAIR
Infarct volume growth | 7 days after stroke onset
  Infarct volume on FLAIR at 7 days minus infarct volume on DWI at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kazunori Toyoda, MD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cerebral and Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Background] Koga M, Toyoda K, Kimura K, Yamamoto H, Sasaki M, Hamasaki T, Kitazono T, Aoki J, Seki K, Homma K, Sato S, Minematsu K; THAWS investigators. THrombolysis for Acute Wake-up and unclear-onset Strokes with alteplase at 0.6 mg/kg (THAWS) Trial. Int J Stroke. 2014 Dec;9(8):1117-24. doi: 10.1111/ijs.12360. Epub 2014 Aug 4. PMID 25088843
- [Background] Toyoda K, Koga M, Hayakawa M, Yamagami H. Acute reperfusion therapy and stroke care in Asia after successful endovascular trials. Stroke. 2015 Jun;46(6):1474-81. doi: 10.1161/STROKEAHA.115.008781. Epub 2015 May 5. PMID 25944322
- [Derived] Toyoda K, Inoue M, Yoshimura S, Yamagami H, Sasaki M, Fukuda-Doi M, Kimura K, Asakura K, Miwa K, Kanzawa T, Ihara M, Kondo R, Shiozawa M, Ohtaki M, Kamiyama K, Itabashi R, Iwama T, Aoki J, Minematsu K, Yamamoto H, Koga M; THAWS trial investigators*. Magnetic Resonance Imaging-Guided Thrombolysis (0.6 mg/kg) Was Beneficial for Unknown Onset Stroke Above a Certain Core Size: THAWS RCT Substudy. Stroke. 2021 Jan;52(1):12-19. doi: 10.1161/STROKEAHA.120.030848. Epub 2020 Dec 10. PMID 33297866
- [Derived] Koga M, Yamamoto H, Inoue M, Asakura K, Aoki J, Hamasaki T, Kanzawa T, Kondo R, Ohtaki M, Itabashi R, Kamiyama K, Iwama T, Nakase T, Yakushiji Y, Igarashi S, Nagakane Y, Takizawa S, Okada Y, Doijiri R, Tsujino A, Ito Y, Ohnishi H, Inoue T, Takagi Y, Hasegawa Y, Shiokawa Y, Sakai N, Osaki M, Uesaka Y, Yoshimura S, Urabe T, Ueda T, Ihara M, Kitazono T, Sasaki M, Oita A, Yoshimura S, Fukuda-Doi M, Miwa K, Kimura K, Minematsu K, Toyoda K; THAWS Trial Investigators. Thrombolysis With Alteplase at 0.6 mg/kg for Stroke With Unknown Time of Onset: A Randomized Controlled Trial. Stroke. 2020 May;51(5):1530-1538. doi: 10.1161/STROKEAHA.119.028127. Epub 2020 Apr 6. PMID 32248771
- See also: THrombolysis for Acute Wake-up and unclear-onset Strokes with alteplase at 0·6 mg/kg (THAWS) Trial — http://onlinelibrary.wiley.com/doi/10.1111/ijs.12360/abstract;jsessionid=763C32F84872E896DA9F27975D7843B6.f01t04